CLINICAL TRIAL: NCT06652724
Title: Relieving Chronic Pain: Psychosomatic Mechanisms and Psychological Interventions in Fibromyalgia and Chronic Headache
Acronym: FIBROMIG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Pavia (Other); Azienda Policlinico Umberto I (Other); Fondazione Mondino (Other); University of Turin, Italy (Other); I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, Federica Galli, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20229NZEKP
Record Dates: First submitted 2024-09-29; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia (FM); Chronic Migraine Headache
Keywords: fibromyalgia; chronic migraine; fmri; psychology; chronic pain; functional magnetic resonance; psychotherapy
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: All participants will be fully aware of the purposes of the research and written informed consent will be obtained from all subjects. All recruited participants will undergo a baseline assessment (T0) using the tests listed in the next section. Patients who meet the inclusion criteria will be enrolled and randomized sequentially into one of three groups: brief psychodynamic therapy (DIT), Expressive Writing Therapy (EST) and controls (TAU). The group selected for the DIT intervention will conduct 16 sessions (one per week) and the group for TSE 8 meetings (one every fortnight) (see description of interventions) for a total intervention time of 4 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic interpersonal therapy (DIT) (Experimental): A total of 54 patients (18 FM, 18 CM, and 18 FibroMig) will receive a brief psychotherapy intervention of 16 sessions (one per week) for a total of 4 months.
  Interventions: Behavioral: Dynamic interpersonal therapy (DIT)
- technique of expressive writing (TSE) (Active Comparator): A total of 54 patients (18 FM, 18 CM, and 18 FibroMig) will receive an expressive writing therapy intervention of 8 meetings (one every fortnight) for a total of 4 months.
  Interventions: Behavioral: technique of expressive writing (TSE)
- treatment as usual (TAU) (Other): A total of 54 patients (18 FM, 18 CM, and 18 FibroMig) will be part of the active control group, planned to monitor specific aspects of the psychotherapeutic intervention, which aims to equate a good standard of primary care.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Dynamic interpersonal therapy (DIT) — Dynamic interpersonal therapy (DIT) is a dynamically oriented brief psychotherapeutic intervention based on attachment and mentalization theory that views symptoms of depression and anxiety as responses to interpersonal difficulties.
  This intervention helps patients to understand the connection between their symptoms and their relationships by identifying a core, non-conscious, repetitive pattern of relating. Previous studies have shown positive results: significant reductions have been observed for the variables somatic symptom severity, depression, anxiety, and general psychiatric symptoms.
  It consists of 16 sessions (one per week) for a total of 4 months.
  Arms: Dynamic interpersonal therapy (DIT)
Behavioral: technique of expressive writing (TSE) — The expressive writing technique created by Pennebaker has shown beneficial health effects in different contexts since, through writing, it is possible to mentally reorganize a difficult event, allowing the mind to find meaning to what has happened or is happening. This technique can be a resource that can promote activation from the ability to recognize, express, and process the unspoken emotional, psychological, and relational, helping to achieve emotional and physiological feedback. Although the application of expressive writing in patients with fibromyalgia is an under-explored area of investigation in the international literature, several studies have shown its effectiveness in some chronic syndromes.
  It consists of 8 meetings (one every fortnight) for a total of 4 months.
  Arms: technique of expressive writing (TSE)
Other: Treatment as Usual (TAU) — The usual treatment involves two contacts by a rheumatologist/neurologist (depending on the clinical condition of the patient) during a four-month period, lasting about 10-15 minutes each, in which patients will be followed up medically. This treatment represents the active control group, planned to monitor specific aspects of the psychotherapeutic intervention, which aims to equate a good standard of primary care.
  Arms: treatment as usual (TAU)

SUMMARY:
Pain is one of the most important manifestations of the disease state and significantly affects people's quality of life. According to the International Association for the Study of Pain (IASP), pain is not only a sensory experience related to the activation of the somato-sensory nervous system, but also an emotional experience, resulting from the cortical and emotional processing of nociceptive signals. This means that perceived pain is the result of a complex interaction between physical sensations and emotional responses.

Pain is classified according to two main criteria: duration and pathophysiological mechanism. In terms of duration, pain can be transient, acute, chronic, or persistent. In terms of pathophysiology, pain can be nociceptive, inflammatory, neuropathic, or nociplastic. The latter, in particular, is characterized by altered nociceptive function, without obvious peripheral damage, and is seen in conditions such as fibromyalgia and chronic migraine.

Chronic pain affects a significant proportion of the population, with estimated prevalence rates between 11% and 40%. According to the US Centers for Disease Control and Prevention, about 20.4 percent of adults suffer from chronic pain. This type of pain is more common in women, people of advanced age, and people with low socioeconomic status. In addition to its physical effects, chronic pain has a major psychological impact, increasing the risk of depression, anxiety, and social isolation. Socially and economically, the costs associated with the treatment and management of chronic pain are high.

Nociplastic pain (DN) refers to a chronic pain state that is not related to visible tissue damage or overt neuropathy, but in which there are alterations in the function of pain sensory pathways. The concept of central sensitization (CS), introduced in the 1990s, describes the amplification of pain signals at the level of the central nervous system, leading to increased sensitivity to pain (hyperalgesia) or pain in response to normally non-painful stimuli (allodynia). This central sensitization has been observed in conditions such as fibromyalgia and chronic migraine.

Fibromyalgia (FM) is a syndrome characterized by widespread musculoskeletal pain associated with fatigue, sleep disturbances, and cognitive deficits. The prevalence of FM is higher among women and tends to be associated with a high level of psychological distress, with anxiety symptoms and depression very common among patients. Although the precise cause of fibromyalgia is still unclear, studies suggest that central sensitization plays a central role in its etiology. Patients with fibromyalgia also have high levels of alexithymia, or the difficulty of identifying and describing emotions, and personality disorders such as avoidant or obsessive-compulsive.

Migraine (CM) affects about 15 percent of the world's population and is characterized by severe headache attacks, often associated with nausea, vomiting, and hypersensitivity to light and sound. Chronic migraine occurs when symptoms occur for at least 15 days per month. Several genetic and environmental factors contribute to the development of migraine, and there is growing evidence indicating a bidirectional relationship between migraine and depression. Anxiety and depression are also risk factors for migraine chronification.

The comorbidity between fibromyalgia and chronic migraine has been the subject of numerous studies. About 45%-80% of patients with fibromyalgia also have migraine, while 20%-36% of patients with migraine also have fibromyalgia. This high incidence of comorbidity suggests that there are common pathophysiological mechanisms between the two conditions, probably related to central sensitization and alterations in nociceptive pain pathways. Recent studies have confirmed that patients with both conditions (FibroMig) may have specific psychological and neurofunctional patterns that distinguish them from those with only one of the two diseases.

This study aims to explore the differences between people with fibromyalgia and chronic migraine, with the goal of identifying distinctive psychological and neurofunctional patterns that could help improve treatments for chronic pain management. An innovative aspect of the project is the identification of the FibroMig sub-population, namely those who suffer from both conditions. These patients might exhibit unique neurophysiological and psychological mechanisms that could be used to develop more targeted treatment strategies.

DETAILED DESCRIPTION:
This research project stems from the intention to observe possible differences between people with FM and CM as clinical conditions representative of diagnostic clusters of DN of a chronic nature, with the ultimate goal of helping to improve treatments for pain management (Cohen, 2022).

The overall goals of the project, in line with the literature review showing a dearth of evidence on mechanisms underlying the onset and maintenance of FM and CM and associated subpopulation (FibroMig), is to identify patterns of psychological and neurofunctional functioning associated with these DN syndromes. In light of the elucidation of such processes that can distinguish these clinical populations, the second general purpose will be to evaluate the efficacy of brief psychodynamic treatments in this area, i.e., to test the efficacy of brief psychodynamic treatment on improvement of pain severity, symptoms of chronic pain pathology, mental pain, psychopathological symptoms (anxiety, depression, etc.), effects on alexithymic functioning and quality of life, in three distinct conditions, FM, CM and comorbidities of FM and CM (FibroMig).

Specifically, the project consists of 2 separate studies that aim to:

* To observe possible differences in psychosocial variables among three groups of patients: isolated form (without comorbidities) of FM, CM and FM and CM comorbidities (FibroMig), compared with a group of healthy subjects (HC) (study 1)
* To evaluate possible differences in the organization of baseline brain functioning (resting-state) between the 3 clinical groups and the healthy control sample (study 1)
* To evaluate the effectiveness of dynamic interpersonal psychotherapy (DIT) on the three patient groups (FM, CM and FibroMig) by comparing them with the application of Expressive Writing Therapy (TSE) and a control group (Treatment as usual - TAU) on improvement with respect to pain severity (VAS), symptom severity (FIQR and symptomatology for CM), mental pain (MPQ), psychopathological symptoms related to anxiety and depression (GAD7, HSRD and PHQ6), level of central sensitization (CSI), level of alexithymia (TAS-20) and Quality of Life (SF-12) (Study 2).

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years;
* at least 5 years of education;
* FM diagnosis according to the criteria reported by Wolfe (2016) for the FM group;
* CM diagnosis according to Olesen (2018) for the CM group;
* medical certification for FM and CM diagnosis for FibroMig group.

Exclusion Criteria:

* severe psychiatric disorders and/or cognitive impairment;
* difficulty understanding/expressing in Italian;
* history of other disorders characterized by chronic pain for FM and CM;
* history of other neurological disorders besides migraine for CM and FibroMig;
* history of other rheumatological disorders besides fibromyalgia for FM and FibroMig;
* For the healthy control group: no diagnosis of FM or CM; no severe psychiatric disorders/cognitive impairment; no or low levels of depression; no history of rheumatological and/or neurological disorders.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
severity of pain | An initial survey at the time of enrollment (T0) then one immediately after the end of the planned interventions (T1, after 4 months of the first one) and finally a survey at 6 months of the end of the intervention (T2).
  To assess the severity of pain, the Visual analogue scales (VAS; Kane, 2005) will be used: it allows pain intensity to be assessed by a ten-point scale with two perpendicular ends: the first end (zero) means no pain, and the second end (ten) means the worst pain.
severity of symptoms | An initial survey at the time of enrollment (T0) then one immediately after the end of the planned interventions (T1, after 4 months of the first one) and finally a survey at 6 months of the end of the intervention (T2).
  To assess symptom severity, the Revised Fibromyalgia Impact Questionnaire (FIQR, Benneet et al., 2009; Salaffi et al., 2013) will be used: it detects the functioning of the person with fibromyalgia by assessing the impairment of functioning and quality of life given by fibromyalgia symptoms.
mental pain | An initial survey at the time of enrollment (T0) then one immediately after the end of the planned interventions (T1, after 4 months of the first one) and finally a survey at 6 months of the end of the intervention (T2).
  To measure mental pain, the Mental Pain Questionnaire (MPQ; Svicher et al., 2019) will be used: it investigates ten aspects of mental pain identified through the literature, namely: presence of mental pain, feeling of helplessness and hopelessness, duration of pain, irreversibility of pain, and intolerance to suffering.
level of central sensitization | An initial survey at the time of enrollment (T0) then one immediately after the end of the planned interventions (T1, after 4 months of the first one) and finally a survey at 6 months of the end of the intervention (T2).
  To measure the level of central sensitization, the Central Sensitivity Inventory (CSI; Chiarotto et al., 2018) will be used: it was developed to assess some psychological symptoms referable to the central sensitivity syndrome. The CSI is intended as a supportive tool to help the clinician identify the presence of the syndrome at the stage of diagnosis that focuses on the person's psychological and emotional experience.
psychopathological symptoms related to anxiety and depression | An initial survey at the time of enrollment (T0) then one immediately after the end of the planned interventions (T1, after 4 months of the first one) and finally a survey at 6 months of the end of the intervention (T2).
  Psychopathological symptoms related to anxiety and depression will be detected using:
  Generalized Anxiety Disorder (GAD-7; Spitzer et al., 2006): for assessing the presence and severity of anxiety symptomatology according to DSM-IV diagnostic criteria Hamilton Depression Rating Scale (HDRS; Hamilton, 1960): for assessing the presence and severity of depressive symptomatology Patient Health Questionnaire (PHQ-9; Kroenke 2001): for assessing the presence and severity of depressive symptomatology according to the DSM-IV diagnostic criteria
alexithymia level | An initial survey at the time of enrollment (T0) then one immediately after the end of the planned interventions (T1, after 4 months of the first one) and finally a survey at 6 months of the end of the intervention (T2).
  To assess the level of alexithymia, the Toronto Alexithymia Scale (TAS-20; Bagby et al., 1994) will be used: this is a self-administered questionnaire consisting of 20 questions that measures difficulty in identifying and describing emotions.
quality of life | An initial survey at the time of enrollment (T0) then one immediately after the end of the planned interventions (T1, after 4 months of the first one) and finally a survey at 6 months of the end of the intervention (T2).
  To measure quality of life, the SF-12 - Quality of Life Assessment (SF-12; Apolone et al., 2001) will be used: this is a generic health survey developed that produces two measures for assessing self-perceived physical and mental health.

SECONDARY OUTCOMES:
traumatic experiences | baseline, pre-intervention
  Traumatic events experienced will be measured with the Traumatic Experiences Checklist (TEC; Nijenhuis et al., 2002): the instrument surveys 29 types of trauma and other potentially overwhelming events: loss of significant others, life-threatening illness or assault, family foster care experience, emotional neglect, emotional abuse, physical abuse, sexual harassment, and sexual trauma
highly sensitivity | baseline, pre-intervention
  To assess highly sensitivity, Highly Sensitive Person Scale (HSP-12 (HSP-12; Aron & Aron, 1997; Lionetti et al., 2018) will be used: investigates the theoretical framework of Sensory Processing Sensitivity, which refers to the innate personal predisposition to wider stimulus processing. In other words, a highly sensitive person is predisposed to perceive external (e.g., auditory, visual) and internal (such as emotions and bodily sensations) sensory stimuli as amplified. The questionnaire specifically assesses the number of details the person is able to perceive from the environment, the intensity with which he or she perceives them, and the threshold of activation.
personality traits | baseline, pre-intervention
  To measure personality traits, the Personality Inventory for DSM-5(PID-5 Short form; Thimm et al., 2016) will be used: it assesses five personality traits, including negative affect, detachment, antagonism, disinhibition, and psychoticism (i.e., the presence of unconventional, strange, eccentric thoughts and behaviors that are not recognized by the home culture).
defensive functioning | baseline, pre-intervention
  To measure defensive functioning, the Defense Mechanism Rating Scales (DMRS-SR-30; Di Giuseppe et al., 2020) will be used: it is an instrument based on the identification of 30 psychological defensive strategies. The DMRS defines each defense mechanism, describes its psychological function, and classifies them into three levels based on functioning (mature, immature, and neurotic).
psychopathological symptoms | baseline, pre-intervention
  The Symptom Checklist-90-Revised (SCL-90-R; Derogatis, 1994) will be used to measure psychopathological symptoms: it assesses psychopathological risk dimensions on 9 dimensions: Somatization, Obsessive-Compulsive Dimension, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, Psychoticism; it also provides a Global Symptom Score (GSI).
reflective function | baseline, pre-intervention
  The Reflective Functioning Questionnaire (RFQ; Fonagy, 2016) will be used to measure reflective function: this is a self-administered questionnaire to assess the ability to think about oneself and others regarding mental states. It provides for two scales, "certainty" indicating hypermentalization, that is, being over-informed about one's own mental states and those of others; and the "uncertainty" scale indicating hypomentalization, that is, showing a total lack of knowledge about mental states and relying on concrete thinking.
attachment style | baseline, pre-intervention
  To measure attachment style, the Relationship Questionnaire (RQ; Bartholomew & Horowitz, 1991) will be used: it assesses attachment style-that is, attitudes and behaviors that contribute to the formation of a specific bond between two people

CONTACTS AND LOCATIONS:
Overall Officials: Federica Galli, Professor, Principal Investigator — University of Roma La Sapienza; Lorys Castelli, Professor, Study Director — University of Turin, Italy; Sara Bottiroli, Professor, Study Director — Università di Pavia; Piercarlo Sarzi-Puttini, MD, Professor, Study Director — University of Milan; Cristina Iannuccelli, Dr, Study Director — Policlinico Umberto I
Locations (2):
- Italy (2):
  - Sapienza University of Rome, Rome, RM
  - Department of Dynamic and Clinical Psychology and Health Studies, Rome, RM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olesen J. International Classification of Headache Disorders. Lancet Neurol. 2018 May;17(5):396-397. doi: 10.1016/S1474-4422(18)30085-1. Epub 2018 Mar 14. No abstract available. PMID 29550365
- [Background] Abbass A, Town J, Holmes H, Luyten P, Cooper A, Russell L, Lumley MA, Schubiner H, Allinson J, Bernier D, De Meulemeester C, Kroenke K, Kisely S. Short-Term Psychodynamic Psychotherapy for Functional Somatic Disorders: A Meta-Analysis of Randomized Controlled Trials. Psychother Psychosom. 2020;89(6):363-370. doi: 10.1159/000507738. Epub 2020 May 19. PMID 32428905
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] Penn IW, Chuang E, Chuang TY, Lin CL, Kao CH. Bidirectional association between migraine and fibromyalgia: retrospective cohort analyses of two populations. BMJ Open. 2019 Apr 8;9(4):e026581. doi: 10.1136/bmjopen-2018-026581. PMID 30962236
- [Background] Nimbi FM, Renzi A, Limoncin E, Bongiovanni SF, Sarzi-Puttini P, Galli F. Central sensitivity in fibromyalgia: testing a model to explain the role of psychological factors on functioning and quality of life. Clin Exp Rheumatol. 2024 Jun;42(6):1187-1197. doi: 10.55563/clinexprheumatol/h8jgv3. Epub 2024 Apr 8. PMID 38607679
- [Background] Kleykamp BA, Ferguson MC, McNicol E, Bixho I, Arnold LM, Edwards RR, Fillingim R, Grol-Prokopczyk H, Turk DC, Dworkin RH. The Prevalence of Psychiatric and Chronic Pain Comorbidities in Fibromyalgia: an ACTTION systematic review. Semin Arthritis Rheum. 2021 Feb;51(1):166-174. doi: 10.1016/j.semarthrit.2020.10.006. Epub 2020 Dec 29. PMID 33383293
- [Background] Karsan N, Goadsby PJ. Migraine Is More Than Just Headache: Is the Link to Chronic Fatigue and Mood Disorders Simply Due to Shared Biological Systems? Front Hum Neurosci. 2021 Jun 3;15:646692. doi: 10.3389/fnhum.2021.646692. eCollection 2021. PMID 34149377
- [Background] Geisser ME, Strader Donnell C, Petzke F, Gracely RH, Clauw DJ, Williams DA. Comorbid somatic symptoms and functional status in patients with fibromyalgia and chronic fatigue syndrome: sensory amplification as a common mechanism. Psychosomatics. 2008 May-Jun;49(3):235-42. doi: 10.1176/appi.psy.49.3.235. PMID 18448779
- [Background] Galli F, Caputi M, Sances G, Vegni E, Bottiroli S, Nappi G, Tassorelli C. Alexithymia in chronic and episodic migraine: a comparative study. J Ment Health. 2017 Jun;26(3):192-196. doi: 10.3109/09638237.2015.1124404. Epub 2016 Jan 6. PMID 26732465
- [Background] Fitzcharles MA, Cohen SP, Clauw DJ, Littlejohn G, Usui C, Hauser W. Nociplastic pain: towards an understanding of prevalent pain conditions. Lancet. 2021 May 29;397(10289):2098-2110. doi: 10.1016/S0140-6736(21)00392-5. PMID 34062144
- [Background] Ferrari MD, Goadsby PJ, Burstein R, Kurth T, Ayata C, Charles A, Ashina M, van den Maagdenberg AMJM, Dodick DW. Migraine. Nat Rev Dis Primers. 2022 Jan 13;8(1):2. doi: 10.1038/s41572-021-00328-4. PMID 35027572
- [Background] de Tommaso M, Sciruicchio V. Migraine and Central Sensitization: Clinical Features, Main Comorbidities and Therapeutic Perspectives. Curr Rheumatol Rev. 2016;12(2):113-26. doi: 10.2174/1573397112666151231110813. PMID 26717950
- [Background] Cho SJ, Perrot S, Sohn JH, Bae JS, Chu MK. Validity and Reliability of the Fibromyalgia Rapid Screening Tool Among Individuals with Chronic Daily Headache: A Clinic-Based Study. Pain Med. 2019 Jun 1;20(6):1193-1201. doi: 10.1093/pm/pny216. PMID 30566656
- [Background] Bottiroli S, Galli F, Viana M, De Icco R, Bitetto V, Allena M, Pazzi S, Sances G, Tassorelli C. Negative Short-Term Outcome of Detoxification Therapy in Chronic Migraine With Medication Overuse Headache: Role for Early Life Traumatic Experiences and Recent Stressful Events. Front Neurol. 2019 Mar 7;10:173. doi: 10.3389/fneur.2019.00173. eCollection 2019. PMID 30899242